CLINICAL TRIAL: NCT03679624
Title: A Phase II Study of Daratumumab Plus Ibrutinib in Patients With Waldenstrӧm's Macroglobulinemia
Brief Title: Daratumumab Plus Ibrutinib in Patients With Waldenstrӧm's Macroglobulinemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry); Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1708018494
Record Dates: First submitted 2018-09-14; First posted 2018-09-20 (Actual); Results first posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-09

CONDITIONS: Waldenstrom Macroglobulinemia; Waldenstrom's Disease; Waldenström; Hypergammaglobulinemia; Waldenstrom's Macroglobulinemia Recurrent; Waldenstrom's Macroglobulinemia of Lymph Nodes; Waldenstrom's Macroglobulinaemia, Without Mention of Remission; Waldenstrom's Macroglobulinemia Refractory
Keywords: treatment naive; relapsed; frontline; refractory; daratumumab; ibrutinib
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Hypergammaglobulinemia; Recurrence | interventions — ibrutinib; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A - Ibrutinib naive (Experimental): Cohort A will consist of subjects who are ibrutinib naïve and appropriate for ibrutinib based treatment. Treatment naïve subjects will be eligible to enroll in this cohort. All subjects in this cohort will receive ibrutinib plus daratumumab
  Interventions: Drug: Ibrutinib; Drug: Daratumumab
- Cohort B - Ibrutinib response plateau (Experimental): Cohort B will consist of subjects who have had at least 6 months of exposure to single agent ibrutinib and who have demonstrated an IgM response plateau defined by two IgM measurements, at least 8 weeks apart that have changed <15% from the previous mark. All subjects in this cohort will receive ibrutinib plus daratumumab
  Interventions: Drug: Ibrutinib; Drug: Daratumumab

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib, 420mg orally, once daily
  Other Names: IMBRUVICA
Drug: Daratumumab — Daratumumab, 16 mg/kg intravenously, weekly for 8 weeks, bi weekly for 16 weeks, then monthly for up to 19 months.
  Other Names: DARZALEX

SUMMARY:
This study evaluates the safety and efficacy of daratumumab in combination with ibrutinib in patients with Waldenstrӧm's macroglobulinemia (WM). The study will evaluate this combination in two cohorts. Cohort A will comprise of ibrutinib naïve WM patients. Patients in this cohort may be treatment naïve or relapsed but who remain ibrutinib naïve. Cohort B will comprise of patients who are currently receiving ibrutinib but whose response to treatment has plateaued. In this cohort, daratumumab will be added on to ibrutinib in an attempt to deepen response.

DETAILED DESCRIPTION:
This is a multi-center, two cohort Phase 2 clinical trial investigating the effectiveness of adding daratumumab to ibrutinib in WM patients. Cohort A will consist of patients who are ibrutinib naïve and appropriate for ibrutinib based treatment. Cohort B will consist of patients who have achieved a response plateau less than a complete remission (CR) on single agent ibrutinib. Subjects in Cohort A will be identified by their treating physician and eligible for enrollment if they are treatment naïve or relapsed after 1 prior therapy for WM and eligible for ibrutinib based treatment.

Subjects in Cohort B will be identified by their treating physician and eligible for enrollment if they have had at least 6 months of exposure to single agent ibrutinib and demonstrate an IgM response plateau defined by two IgM measurements, at least 8 weeks apart that have changed <15% from the previous mark. In Cohort B response assessment will be measured from initial IgM level prior to ibrutinib initiation.

Enrolled subjects will be prescribed commercial ibrutinib, 420mg PO daily. The investigational agent, daratumumab will be administered based on FDA approved dosing in multiple myeloma (16mg/kg) with 8 weekly induction treatments during Cycles 1 and 2, followed by every other week dosing for Cycles 3-6, then monthly dosing from Cycle 7 until Cycle 25 at which point subjects will continue with ibrutinib as monotherapy until Cycle 52 (4 years total) which is the predefined study completion for enrolled subjects at which point they will complete follow-up. Study visits and response assessments with IgM measurements will occur with each cycle for the first year then every three cycles after cycle 13. Subjects with measureable extramedullary disease will have CT scans every 6 cycles until radiographic CR. Patients will be considered evaluable for response if they completed the initial 8 weeks of daratumumab induction therapy and evaluable for toxicity if receiving one dose of daratumumab. Patients will continue on combination therapy for 2 years or until disease progression or unacceptable toxicities at which point subjects will come off trial. Patients achieving a CR after two years of combination therapy will be given an option to continue with single agent commercial ibrutinib.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a diagnosis of WM and meet the requirements for active therapy as defined by the 2nd International Workshop on Waldenstrom's Macroglobulinemia
* Age ≥18 years of age
* Ibrutinib naïve or previously treated patients currently on ibrutinib with a plateau in disease response are eligible to participate.

  1. Ibrutinib naïve subjects may be either treatment naïve or previously treated but ibrutinib naïve to enter cohort A.
  2. Subjects entering cohort B must have a plateau response on ibrutinib defined as ≥ 6 months of ibrutinib treatment with 2 IgM measurements at least 2 months apart with ≤ 15% change from the previous measurement. Subjects with IgM level < 0.7 g/dL will be eligible if their IgM level increases < 0.15 g/dL over two subsequent IgM measurements as defined above.
* Subjects must have measurable disease defined by a serum IgM level ≥0.5g/dL
* Eastern Cooperative Oncology Group performance status of 0-2
* Hematology values must be within the following limits:

  1. Absolute neutrophil count (ANC) ≥ 1000/mm3 independent of growth factor support for 7 days of study entry if cytopenias are due to marrow involvement.
  2. Platelets ≥ 50,000/mm3 independent of transfusion support within 7 days of study entry. TPO mimetics are not allowed to meet eligibility criteria.
  3. Hemoglobin ≥ 8g/dL, independent of transfusion support within 7 days of study entry
* Biochemical values within the following limits:

  d. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x upper limit of normal (ULN)

  e. Total bilirubin ≤ 2 x ULN unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin

  f. Creatinine clearance (CLcr) > 25 ml/min
* Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. Men must agree to not donate sperm during and after the study. For females, these restrictions apply for 1 month after the last dose of study drug. For males, these restrictions apply for 3 months after the last dose of study drug.
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin (beta-hCG) or urine beta hCG pregnancy test at Screening. Women who are pregnant or breastfeeding are ineligible for this study.
* Subjects must be able to sign (or their legally-acceptable representatives must sign) an informed consent indicating that they understand the rational of the study and can participate in all study procedures.

Exclusion Criteria:

* Subject does not have a recorded IgM level recorded within 3 months prior to ibrutinib initiation.
* Subject meeting definition of disease progression while on ibrutinib. Subjects with IgM levels < 0.7gdL are given special consideration. Please see inclusion criteria for 2b.
* Subjects in cohort B experiencing ongoing non hematologic toxicities attributable to ibrutinib > Grade 1 will be excluded from study entry.
* Major surgery or a wound that has not fully healed within 4 weeks of enrollment.
* Evidence of disease transformation at time of enrollment.
* Waldenstrom's complicated by amyloidosis
* Known central nervous system lymphoma.
* History of stroke or intracranial hemorrhage within 6 months prior to randomization.
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists (eg, phenprocoumon).
* Requires chronic treatment with strong CYP3A inhibitors. Subjects that required strong CYP3A inhibitors but completed a course of treatment can be considered for enrollment after a washout period of 14 days prior to study drug administration.
* Requires strong CYP3A inducers. Subjects that required strong CYP3A inducers but completed a course of treatment can be considered for enrollment after a washout period of 14 days prior to study drug administration.
* Patients with history of Chronic Obstructive Pulmonary Disease or Reactive Airway disease must have PFTs with FEV1 calculated. Patients with a FEV1 ≤ 50% of predicted normal will be excluded.
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification.
* Vaccinated with live, attenuated vaccines within 4 weeks of randomization.
* Seropositive for human immunodeficiency virus (HIV).
* Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (i.e., subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
* Seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy).
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk.
* Active malignancy not treated with curative intent within 2 years of study entry. Nonmelanotic skin cancers and cervical carcinoma in situ are excluded from this criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John N. Allan, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: WCM Joint Clinical Trials Office — https://jcto.weill.cornell.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort A - Ibrutinib Naive | Cohort B - Ibrutinib Response Plateau
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: 0 subjects were enrolled in Cohort B.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A - Ibrutinib Naive | Cohort B - Ibrutinib Response Plateau | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 1 |  | 1
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety of Combination Treatment With Ibrutinib and Daratumumab as Measured by the Number of Patients That Experience 1 or More Adverse Event
Description: Number of patients that experience 1 or more adverse event
Time Frame: 3 months
Population: 0 subjects were enrolled in Cohort B.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A - Ibrutinib Naive | Cohort B - Ibrutinib Response Plateau
Number analyzed (Participants) | 1 | 0
Participants | 1 |

2. Secondary Outcome: Major Response Rate in Cohort A
Description: Number of patients in Cohort A who achieve VGPR, PR, or CR
Time Frame: 5 years
Population: The patient in Cohort A did not complete enough cycles to evaluate for a response. 0 subjects were enrolled in Cohort B.
Arm/Group | Cohort A - Ibrutinib Naive | Cohort B - Ibrutinib Response Plateau
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Deepening of Response Rate in Cohort B After Daratumumab Addition
Description: Number of patients in Cohort B who achieve a VGPR, PR, or CR from baseline IgM prior to ibrutinib
Time Frame: 5 years
Population: The patient in Cohort A did not complete enough cycles to evaluate for a response. 0 subjects were enrolled in Cohort B.
Arm/Group | Cohort A - Ibrutinib Naive | Cohort B - Ibrutinib Response Plateau
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Duration of Response
Description: Measured from time of first response to progression or death, measured in months.
Time Frame: 5 years
Population: The patient in Cohort A did not complete enough cycles to evaluate for a response. 0 subjects were enrolled in Cohort B.
Arm/Group | Cohort A - Ibrutinib Naive | Cohort B - Ibrutinib Response Plateau
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to Progression
Description: Measured from time of study drug administration to progression, measured in months.
Time Frame: 5 years
Population: Cohort A participant did not complete enough cycles to get a response. 0 subjects were enrolled in Cohort B.
Arm/Group | Cohort A - Ibrutinib Naive | Cohort B - Ibrutinib Response Plateau
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Progression Free Survival
Description: Measured from time of study drug administration to progression or death, measured in months.
Time Frame: 3 months
Population: Cohort A participant did not complete enough cycles to evaluate for response. 0 subjects were enrolled in Cohort B.
Measure: Median (Standard Deviation); unit: months
Arm/Group | Cohort A - Ibrutinib Naive | Cohort B - Ibrutinib Response Plateau
Number analyzed (Participants) | 1 | 0
months | NA — lack of participants with events |

7. Secondary Outcome: Overall Survival
Description: Measured from time of study drug administration to death, measured in months.
Time Frame: 3 months
Population: The patient in Cohort A did not complete enough cycles to evaluate for a response. 0 subjects were enrolled in Cohort B.
Measure: Median (Standard Deviation); unit: months
Arm/Group | Cohort A - Ibrutinib Naive | Cohort B - Ibrutinib Response Plateau
Number analyzed (Participants) | 1 | 0
months | NA — lack of participants with events |

ADVERSE EVENTS:
Time Frame: 3 months
Description: 0 subjects were enrolled in Cohort B
Arm/Group | Cohort A - Ibrutinib Naive | Cohort B - Ibrutinib Response Plateau
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A - Ibrutinib Naive (N=1) | Cohort B - Ibrutinib Response Plateau (N=0)
Elevated ALT/AST (General disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A - Ibrutinib Naive (N=1) | Cohort B - Ibrutinib Response Plateau (N=0)
Vomiting (Metabolism and nutrition disorders) | 1 (1) | 0 — grade 1
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infusion related (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Infusion-related reaction
Scratchy Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ALT increased (Investigations) | 1 (1) | 0 (0)
AST increased (Investigations) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Malaise- flu like symptoms (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/24/NCT03679624/Prot_SAP_000.pdf